CLINICAL TRIAL: NCT01286779
Title: BAX 326 (Recombinant Factor IX): Evaluation of Safety, Immunogenicity, and Hemostatic Efficacy in Previously Treated Patients With Severe (FIX Level < 1%) or Moderately Severe (FIX Level <= 2%) Hemophilia B - A Continuation Study
Brief Title: BAX 326 (rFIX) Continuation Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 251001; 2010-022726-33 (EudraCT Number)
Record Dates: First submitted 2011-01-26; First posted 2011-01-31 (Estimated); Results first posted 2018-09-10 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-04

CONDITIONS: Hemophilia B
MeSH Terms: conditions — Hemophilia B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BAX 326 (Experimental)
  Interventions: Biological: BAX 326 (Recombinant factor IX)

INTERVENTIONS:
Biological: BAX 326 (Recombinant factor IX) — The treatment with BAX 326 will be at the discretion of the investigator and will consist of either twice weekly prophylactic treatment with 50 IU/kg, modified prophylaxis, or on-demand treatment.

SUMMARY:
The purpose of this BAX 326 Continuation Study is to further investigate incremental recovery over time, the hemostatic efficacy, the safety, immunogenicity, and health-related quality of life (HR QoL) of BAX 326 in previously treated patients (PTPs) with severe and moderately severe hemophilia B who participated in BAX 326 pivotal study 250901 or BAX 326 pediatric study 251101.

ELIGIBILITY:
Main Inclusion Criteria:

* Subject and/or legal representative has/have voluntarily provided signed informed consent
* Subject has completed Baxter clinical study 250901 (pivotal study) or Baxter clinical study 251101 (pediatric study)
* Subject was 12 to 65 years old at the time of screening for Study 250901 or < 12 years old at the time of screening for Study 251101
* Subject has severe (FIX level < 1%) or moderately severe (FIX level 1-2%) hemophilia B (based on the one stage activated partial thromboplastin time (aPTT) assay), as tested at screening at the central laboratory
* Subject has not developed an inhibitory FIX antibody during Baxter Pivotal Study 250901 or Pediatric Study 251101

Main Exclusion Criteria:

* Subject received factor IX product(s) other than BAX 326 upon completion of Baxter Pivotal Study 250901 or Pediatric Study 251101
* Subject has been diagnosed with an acquired hemostatic defect other than hemophilia B
* For subjects transferring from Pivotal Study 250901: Subject's weight is < 35 kg or > 120 kg
* Subject is planned to take part in any other clinical study, with the exception of BAX 326 Surgery study as described in this protocol, during the course of the Continuation Study

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2011-04-12 (Actual); Primary Completion 2017-06-29 (Actual); Study Completion 2017-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (42):
- Instituto de Hematología y Medicina Clíncia Rubén Dávoli, Rosario, Argentina
- UNIFESP - Universidade Estadual de Sao Paulo, São Paulo, Brazil
- Specialized Haematological Hospital "Joan Pavel", Sofia, Bulgaria
- Hospital Dr. Sotero del Rio, Santiago, Chile
- Colombia (3):
  - Hospital de San Jose, Bogotá
  - Centro Medico Imbanaco, Cali
  - Hospital Pablo Tobon Uribe, Medellín
- Klinika detské hematologie a onkologie, Prague, Czechia
- Maulana Azad Medical College and Associated Hospital, New Delhi, India
- St. James's Hospital, National Center for Hereditary Coagulation Disorders, Dublin, Ireland
- Italy (5):
  - University Hospital Policlinico Vittorio Emanuele, Hospital Ferrarotto Alessi, Catania
  - University Hospital Careggi, Agency of Hemophilia - Regional Reference Center for Inherited Bleeding, Florence
  - University of Foggia Riuniti Hospital, Department of Clinical and Experimental Medicine, Foggia
  - Hospital San Giovanni Bosco, Center for Hemophilia and Thrombosis, Department of Hematology, Naples
  - Padova University Hospital, Medical Clinic II, Center for Hemophilia, Padua
- Japan (3):
  - Nara Medical University, Department of Pediatrics, Nara
  - Tokyo Medical University, Tokyo
  - Ogikubo Hospital, Tokyo
- Poland (7):
  - Hematology and Transplantology Clinic, University Clinic Centre - Medical University Hospital, Gdansk
  - University Pediatric Hospital in Cracow, Krakow
  - Medical College of the Jagiellonian University, Department of Hematology, Krakow
  - Copernicus Hospital, Medical University in Lodz, Department of Hematology, Lodz
  - Professor Tadeusz Sokolowski Independent Public Teaching Hospital No. 1 of the Pomeranian Medical University in Szczecin, Szczecin
  - Klinika Hematologii, Warsaw
  - Institute of Haematology and Transfusion Medicine, Warsaw
- Romania (2):
  - Prof. Dr. C.T. Nicolau National Institute for Transfusional Hematology, Bucharest
  - Louis Turcanu Emergency Clinical Children´s Hospital, Timișoara
- Russia (5):
  - Federal State Institution Kirov Hematology and Blood Transfusion Research Institute under the Federal Agency for High-Tech Medical Care, Kirov
  - Pediatric Regional Clinical Hospital, Hematology Department, Krasnodar
  - Hematology Research Center RAMS, Department of Reconstructive Orthopedics for Haemophilia Patients, Moscow
  - Republican Center for Hemophilia Treatment Outpatient Clinic No. 37, Saint Petersburg
  - Regional clinical hospital, Yekaterinburg
- Malmö University Hospital, Department of Coagulation Disorders, Malmo, Sweden
- Taiwan (6):
  - Taipei Medical University Hospital, Taipei City, Taipei
  - Chung-Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Tri-Service General Hospital, Taipei
- State Institution "Institute of Blood Pathology and Transfusion Medicine of the Academy of Medical Sciences of Ukraine", Lviv, Ukraine
- United Kingdom (2):
  - Katharine Dormandy Haemophilia Centre and Haemostasis Unit, Royal Free Hospital, London
  - Manchester Children's Hospital, Manchester

REFERENCES:
- [Derived] Windyga J, Stasyshyn O, Lissitchkov T, Mamonov V, Serban M, Rusen L, Ploder B, Tangada S. Safety, Immunogenicity, and Hemostatic Efficacy of Nonacog Gamma in Patients With Severe or Moderately Severe Hemophilia B: A Continuation Study. Clin Appl Thromb Hemost. 2020 Jan-Dec;26:1076029620950836. doi: 10.1177/1076029620950836. PMID 32866032

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment was conducted at 40 clinical sites in 18 countries. A total of 117 participants were enrolled. Of these, 65 participants transitioned from BAX326 pivotal study, 20 participants transitioned from BAX326 pediatric study and 32 participants were newly recruited.
Pre-assignment Details: Of 117 enrolled participants, 115 received treatment with IP. All 85 participants who transitioned from the pivotal/pediatric studies continued to receive IP in this study. Of the 32 newly recruited participants, 30 received treatment with IP. 1 participant did not meet the entry criteria and 1 participant discontinued the study prior treatment.
Groups:
- BAX 326: Participants treated with BAX 326
Period: Overall Study
Arm/Group | BAX 326
Started | 115
Completed | 96
Not Completed | 19
Not completed — Withdrawal by Subject | 9
Not completed — Protocol Violation | 5
Not completed — Physician Decision | 2
Not completed — Participant had scheduled surgery | 1
Not completed — Participant moved to another country | 1
Not completed — Discontinued by sponsor | 1

BASELINE CHARACTERISTICS:
Arm/Group | BAX 326
Number analyzed (Participants) | 115
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.6 (16.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 115
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 99
  Race: Black or African American | 1
  Race: Asian | 10
  Race: Other | 5

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events Possibly or Probably Related to the Investigational Product
Description: Possibly or probably related adverse events that occurred during or after first BAX326 infusion.
Time Frame: Assessed (based on patient diary) every 3 months until study completion (when BAX326 is licensed in the respective country or the participant has accumulated approximately 100 exposure days to BAX 326, whichever is last).
Measure: Number; unit: Adverse Events
Arm/Group | BAX 326
Number analyzed (Participants) | 115
Adverse Events | 2

2. Secondary Outcome: Treatment of Bleeding Episodes: Number of Infusions Per Bleeding Episode Required Until Bleed Resolution
Description: Number of Infusions of BAX326 that were required until bleed resolution.
Time Frame: Throughout the study from screening to study completion (when BAX326 is licensed in the respective country or the participant has accumulated approximately 100 exposure days to BAX 326, whichever is last).
Population: Only bleeding episodes that were exclusively treated with BAX 326 are considered.
Measure: Mean (Standard Deviation); unit: Number of infusions
Units Other Than Participants: Bleeding episodes
Groups:
- Standard Prophylaxis: Participants treated with BAX 326 with twice weekly prophylactic infusions of 50 IU/kg
- Modified Prophylaxis: Participants treated with BAX 326 with prophylactic treatment determined by the investigator. The dose could be increased up to 100 IU/kg if indicated.
- PK Tailored Prophylaxis: Participants treated with BAX 326 with PK tailored prophylaxis base on participant's individual PK with maximum dose of 120 IU/kg.
- Overall Prophylaxis: All participants who received BAX 326 as prophylactic regimen (standard prophylaxis, modified prophylaxis and PK-tailored prophylaxis)
- On-Demand: All participants who received BAX 326 as on-demand regimen.
Arm/Group | BAX 326 | Standard Prophylaxis | Modified Prophylaxis | PK Tailored Prophylaxis | Overall Prophylaxis | On-Demand
Number analyzed (Participants) | 115 | 108 | 26 | 3 | 110 | 13
Number analyzed (Bleeding episodes) | 1112 | 542 | 108 | 8 | 658 | 454
Number of infusions | 1.8 (1.65) | 2.1 (2.12) | 1.9 (1.41) | 1.3 (0.46) | 2.0 (2.01) | 1.5 (0.79)

3. Secondary Outcome: Treatment of Bleeding Episodes: Overall Hemostatic Efficacy Rating at Resolution of Bleed
Description: Overall clinical efficacy rating of bleeding episodes was done at resolution of bleed according these rating scale: Excellent=Full relief of pain and cessation of objective signs of bleeding after a single infusion. No additional infusion is required for the control of bleeding. Administration of further infusion would not affect the scoring. Good=Definite pain relief and/or improvement in signs of bleeding after a single infusion. Possibly requires more than 1 infusion for complete resolution. Fair=Probable and/or slight relief of pain and slight improvement in signs of bleeding after a single infusion. Required more than 1 infusion for complete resolution. None=No improvement or condition worsens.
Time Frame: as for outcome 2
Population: Only bleeding episodes that were exclusively treated with BAX 326 are considered.
Measure: Number; unit: Number of infusions
Units Other Than Participants: Bleeding Episodes
Arm/Group | BAX 326 | Standard Prophylaxis | Modified Prophylaxis | PK Tailored Prophylaxis | Overall Prophylaxis | On-Demand
Number analyzed (Participants) | 115 | 108 | 26 | 3 | 110 | 13
Number analyzed (Bleeding Episodes) | 1112 | 542 | 108 | 8 | 658 | 454
Number of infusions
  Excellent | 341 | 168 | 51 | 0 | 219 | 122
  Good | 650 | 281 | 40 | 0 | 321 | 329
  Fair | 115 | 90 | 17 | 6 | 113 | 2
  None | 6 | 3 | 0 | 2 | 5 | 1

4. Secondary Outcome: Annualized Bleed Rate During Prophylaxis Treatment
Description: Annualized bleed rate (ABR) was calculated as (number of bleeding episodes/observed treatment period in days)*365.25
Time Frame: For prophylactic treatment the period from first to last prophylactic infusion is considered.
Population: Only participants with an observation period of at least 3 months with BAX326 on prophylactic treatment were included in the analysis.
Measure: Median (Full Range); unit: Bleeds per year
Arm/Group | Standard Prophylaxis | Modified Prophylaxis | PK Tailored Prophylaxis | Overall Prophylaxis
Number analyzed (Participants) | 106 | 22 | 2 | 108
Bleeds per year | 1.3 [0.0 to 78.7] | 1.4 [0.0 to 34.6] | 1.9 [0.5 to 3.3] | 1.3 [0.0 to 52.2]

5. Secondary Outcome: Consumption of BAX 326: Number of Infusions Per Month and Per Year
Description: The number of infusions consumed per month and per year for the prophylactic and on-demand treatment regimens.
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: Number of infusions
Arm/Group | Standard Prophylaxis | Modified Prophylaxis | PK Tailored Prophylaxis | Overall Prophylaxis | On-Demand
Number analyzed (Participants) | 108 | 26 | 3 | 110 | 13
Number of infusions
  Number of infusions per month | 8.5 (1.25) | 10.8 (4.34) | 4.0 (0.60) | 8.4 (1.38) | 3.6 (2.44)
  Number of infusions per year | 101.8 (15.03) | 130.2 (52.13) | 48.3 (7.23) | 101.1 (16.50) | 43.1 (29.28)

6. Secondary Outcome: Consumption of BAX 326: Weight Adjusted Consumption Per Month and Per Year
Description: The weight adjusted consumption of BAX 326 per month and per year for the prophylactic and on-demand treatment regimens.
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: IU/kg
Arm/Group | Standard Prophylaxis | Modified Prophylaxis | PK Tailored Prophylaxis | Overall Prophylaxis | On-Demand
Number analyzed (Participants) | 108 | 26 | 3 | 110 | 13
IU/kg
  Weight adjusted BAX 326 consumption per month | 462.3 (102.05) | 684.4 (337.70) | 250.9 (41.37) | 464.2 (111.46) | 199.8 (124.18)
  Weight adjusted BAX 326 consumption per year | 5547.8 (1224.65) | 8212.4 (4052.36) | 3010.3 (496.44) | 5570.7 (1337.53) | 2397.4 (1490.22)

7. Secondary Outcome: Consumption of BAX326: Weight Adjusted Consumption Per Bleeding Episode
Description: The weight adjusted consumption of BAX 326 per bleeding episode for the prophylactic and on-demand treatment regimens. Only infusions required until the resolution of bleed are considered.
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: IU/kg
Units Other Than Participants: Bleeding episodes
Arm/Group | Standard Prophylaxis | Modified Prophylaxis | PK Tailored Prophylaxis | Overall Prophylaxis | On-Demand
Number analyzed (Participants) | 108 | 26 | 3 | 110 | 13
Number analyzed (Bleeding episodes) | 542 | 109 | 8 | 659 | 453
IU/kg | 124.2 (140.70) | 114.8 (99.41) | 67.4 (34.39) | 122.0 (134.02) | 82.6 (48.21)

8. Secondary Outcome: Development of Inhibitory and Total Binding Antibodies to Factor IX
Description: Testing for inhibitory and total binding antibodies to Factor IX (FIX). Development during study means negative at screening and positive at any subsequent visit. Treatment emergent means more than 2-dilution increase as compared to the pre-study titer at screening.
Time Frame: Laboratory assessment for immunology were done at screening, at exposure day 1, at week 4 (± 1 week), at month 3 (±1 week), thereafter, every 3 months (± 1 week) and at study completion/termination.
Measure: Count of Participants; unit: Participants
Arm/Group | BAX 326
Number analyzed (Participants) | 115
Participants
  Inhibitory antibodies to FIX-develop. during study | 0
  Inhibitory antibodies to FIX-treatment emergent | 0
  Total bind. antibodies to FIX-develop.during study | 0
  Total binding antibodies to FIX-treatment emergent | 0

9. Secondary Outcome: Development of Antibodies to Chinese Hamster Ovary Proteins (CHO Proteins) and rFurin
Description: Testing for antibodies to CHO proteins and rFurin. Development during study means negative at screening and positive at any subsequent visit. Treatment emergent means more than 2-dilution increase as compared to the pre-study titer at screening.
Time Frame: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | BAX 326
Number analyzed (Participants) | 115
Participants
  Antibodies to CHO - developed during study | 0
  Antibodies to CHO - treatment emergent | 0
  Antibodies to rFurin - developed during study | 4
  Antibodies to rFurin - treatment emergent | 4

10. Secondary Outcome: Occurrence of Severe Allergic Reactions and Thrombotic Events
Description: The occurrence of severe allergic reactions and thrombotic events was assessed.
Time Frame: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | BAX 326
Number analyzed (Participants) | 115
Participants
  Severe allergic reactions | 0
  Thrombotic events | 0

11. Secondary Outcome: Clinical Significant Changes in Routine Laboratory Parameters and Vital Signs
Description: Hematology panel consists of complete blood count (hemoglobin, hematocrit, erythrocytes, leukocytes) with differential (ie, basophils, eosinophils, lymphocytes, monocytes, neutrophils), mean corpuscular volume, mean corpuscular hemoglobin concentration and platelet count. Clinical chemistry panel consists of sodium, potassium, chloride, bicarbonate, total protein, albumin, alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin, alkaline phosphatase, blood urea nitrogen, creatinine and glucose. Vital signs include body temperature, respiratory rate, pulse rate, supine systolic and diastolic blood pressure. CS=clinically significant, NCS=not clinically significant. Change from Screening to End of Study is reported.
Time Frame: Measurements at screening and at study completion/termination are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | BAX 326
Number analyzed (Participants) | 115
Participants
  Hematology: Change from normal to abnormal CS | 2
  Hematology:Change from abnormal NCS to abnormal CS | 1
  Chemistry: Change from normal to abnormal, CS | 1
  Chemistry: Change from abnormal NCS to abnormal CS | 3
  Change in vital signs | 0

12. Secondary Outcome: Pharmacokinetics: Incremental Recovery (IR) Over Time
Description: PK infusion with investigational product was administered after a wash out period of at least 5 days. Incremental recovery is calculated as IR30min = (C30min [IU/dL] - Cpre-infusion [IU/dL]) / dose per kg body weight [IU/kg] where C30min and Cpre-infusion relate to the unadjusted concentration values.
Time Frame: IR over time was measured as Baseline and at Completion/Termination visit within 30 minutes pre-infusion and at 30 (± 5) minutes post-infusion.
Population: Analysis was done on all participants who received investigational product. All cases with a dosage higher than 120 IU/kg were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: (IU/dL):(IU/kg)
Arm/Group | BAX 326
Number analyzed (Participants) | 115
(IU/dL):(IU/kg)
  Baseline: number analyzed (Participants) | 110
  Baseline | 0.85 (0.207)
  End of Study: number analyzed (Participants) | 108
  End of Study | 0.85 (0.286)
  Change from baseline to end of study: number analyzed (Participants) | 104
  Change from baseline to end of study | -0.005 (0.259)

13. Secondary Outcome: Pharmacokinetics: Area Under the Plasma Concentration Versus Time Curve From Time 0 to Infinity (AUC 0-∞)
Description: After a wash out period of at least 5 days PK infusion with investigational product was administered. AUC 0-∞ is defined as AUC 0-t + Ct/lambda z, where t is the time of last quantifiable concentration, Ct is the last quantifiable concentration.
Time Frame: PK assessments were done within 30 minutes pre-infusion and post-infusion at 30 (± 5) minutes, 9 hours (± 30 minutes), 24 (± 2) hours, 48 (± 2) hours and 72 (± 2) hours
Population: The pharmacokinetic analysis set comprises all participants who underwent an abbreviated PK study.
Measure: Mean (Standard Deviation); unit: IU*hr/dL
Arm/Group | BAX 326
Number analyzed (Participants) | 6
IU*hr/dL | 1335.56 (299.83)

14. Secondary Outcome: Pharmacokinetics: Elimination Phase Half-life (T1/2)
Description: PK infusion with investigational product was administered after a wash out period of at least 5 days. Elimination phase half-life is calculated as T1/2=log e (2) / lambda z where the elimination rate constant (lambda z) will be obtained by log e - linear fitting using least squares deviation to at least the last 3 quantifiable concentrations above pre-infusion level.
Time Frame: as for outcome 13
Population: The pharmacokinetic analysis set comprises all participants who underwent an abbreviated PK study.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | BAX 326
Number analyzed (Participants) | 6
hours | 28.52 (4.12)

15. Secondary Outcome: Pharmacokinetics: Mean Residence Time (MRT)
Description: PK infusion with investigational product was administered after a wash out period of at least 5 days. Mean residence time is calculated as total area under the moment curve divided by the total area under the curve. MRT=(AUMC0-∞[h2*IU/dL])/(AUC0-∞[h*IU/dL]) - TI/2 where AUMC0-∞ is determined in a similar manner as AUC0-∞ and TI represents infusion duration in hours.
Time Frame: as for outcome 13
Population: The pharmacokinetic analysis set comprises all participants who underwent an abbreviated PK study.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | BAX 326
Number analyzed (Participants) | 6
hours | 29.97 (2.72)

16. Secondary Outcome: Pharmacokinetics: Systemic Clearance (CL)
Description: PK infusion with investigational product was administered after a wash out period of at least 5 days. Systemic clearance is balculated as the dose in IU/kg divided by the total AUC. CL= Dose[IU/kg] / AUC0-∞[h*IU/dL]
Time Frame: as for outcome 13
Population: The pharmacokinetic analysis set comprises all participants who underwent an abbreviated PK study.
Measure: Mean (Standard Deviation); unit: dL/kg/hours
Arm/Group | BAX 326
Number analyzed (Participants) | 6
dL/kg/hours | 0.06 (0.014)

17. Secondary Outcome: Pharmacokinetics: Volume of Distribution at Steady State (Vss)
Description: PK infusion with investigational product was administered after a wash out period of at least 5 days. Apparent steady state volume of distribution is calculated as Vss = CL * MRT CL=Systemic Clearance and MRT=Mean residence time
Time Frame: as for outcome 13
Population: The pharmacokinetic analysis set comprises all participants who underwent an abbreviated PK study.
Measure: Mean (Standard Deviation); unit: dL/kg
Arm/Group | BAX 326
Number analyzed (Participants) | 6
dL/kg | 1.78 (0.42)

18. Secondary Outcome: Pharmacokinetics: Incremental Recovery (IR)
Description: as for outcome 12
Time Frame: as for outcome 13
Population: The pharmacokinetic analysis set comprises all participants who underwent an abbreviated PK study.
Measure: Mean (Standard Deviation); unit: (IU/dL):(IU/kg)
Arm/Group | BAX 326
Number analyzed (Participants) | 6
(IU/dL):(IU/kg) | 0.85 (0.196)

19. Secondary Outcome: Changes in Health Related Quality of Life (HR QoL) Based on Questionnaire SF-36
Description: The Short Form (36) Health Survey (SF-36) is a 36-item validated, generic HR QoL instrument suitable for participants of 17 years of age or older. The SF-36 consists of eight scaled scores (vitality, physical functioning, bodily pain, general health, mental health, physical role functioning, emotional role functioning, social role functioning) which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability. The mental health component summary score ranged from 19.5 to 64.2 with higher scores indicating less disability. The physical health component summary scores ranged from 18.6 to 59.6 with higher scores indicating less disability.
Time Frame: Baseline at exposure day 1 and at study completion/termination.
Population: Only newly recruited participants are included as baseline values were not reported for transitioning participants. Only subjects how received prophylaxis treatment are included.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | BAX 326
Number analyzed (Participants) | 24
Score on a scale
  SF-36 Bodily Pain | 6.7 (12.66)
  SF-36 General Health | 3.2 (9.32)
  SF-36 Mental Health | 0.7 (14.72)
  SF-36 Mental Health Component Score | 0.8 (12.08)
  SF-36 Physical Functioning | 4.2 (10.46)
  SF-36 Physical Health Component Score | 5.7 (8.43)
  SF-36 Role-Emotional | 2.3 (11.57)
  SF-36 Role-Physical | 4.5 (10.28)
  SF-36 Social Functioning | 4.5 (11.67)
  SF-36 Vitality | 2.0 (8.87)

20. Secondary Outcome: Changes in Health Related Quality of Life Using the Peds QL
Description: The Pediatric Quality of Life Inventory (Peds QL) is a generic health related quality of life instrument designed specifically for a pediatric population and captures following domains: physical functioning, emotional functioning, social functioning and school functioning. The Peds-QL total score consist of all 23 items of all domains. Score range from 0-100 and higher scores indicate better quality of life (collected scores ranged from 44.6 to 98.9). The Peds-QL Physical Health Summary score consists of 8 items from the physical functioning domain. Score range from 0-100 and higher scores indicate better quality of life (collected scores ranged from 40.6 to 100.0) The Psychosocial Health Summary score consists of 15 items from the emotional, social and school functioning domains. Score range from 0 to 100 and higher scores indicate better quality of life (collected scores ranged from 46.7 to 100.0).
Time Frame: Baseline at exposure day 1 and at study completion/termination.
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | BAX 326
Number analyzed (Participants) | 4
Score on a scale
  Peds-QL Physical Health Summary Score | -2.3 (18.47)
  Peds-QL Psychosocial Health Summary Score | 3.8 (5.99)
  Peds-QL Total Score | 1.6 (10.14)

21. Secondary Outcome: Changes in Health Related Quality of Life (HR QoL) Based on Questionnaire Haemo-QoL and Haem-A-QoL
Description: The Hemophilia Quality of Life Questionnaire (Haemo-QoL) and the Hemophilia Quality of Life Questionnaire for Adults (Haem-A-Qol) instruments have been developed and used in hemophilia A patients. As a hemophilia-specific instrument, this measure assesses very specific aspects of dealing with hemophilia. The areas covered by this instrument are: physical health, sports/leisure, school/work, dealing with hemophilia, and outlook for the future. Haemo-QoL is used for participants aged 8 to 16 years and total scores range from 0 to 100 with higher scores indicating low quality of life (collected scores ranged from 0.0 to 44.3) Haem-A-QoL is used for participants aged 17 years and older and total scores range from 0 to 100 with higher scores indicating low quality of life (collected scores ranged from 4.9 to 76.8).
Time Frame: Baseline at exposure day 1 and at study completion/termination.
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | BAX 326
Number analyzed (Participants) | 16
Score on a scale
  Haem-A-QoL Total Score | -3.0 (9.45)
  Haemo-QoL Total Score: number analyzed (Participants) | 1
  Haemo-QoL Total Score | -0.7 (NA) — only 1 participant analyzed

22. Secondary Outcome: Changes in Health Related Quality of Life (HR QoL) Based on Questionnaire EQ-5D and Pain Score.
Description: The EQ-5D captures overall HR QoL (phyiscal, mental and social functioning). A health utility score can be calculated from this measure, adult and proxy versions available. EQ-5D Visual Analog Scale (EQ-5D VAS):Respondents specify their level of agreement to a statement by indicating a position along a continuous line between two endpoints (scale range from 0 to 100). Score 0 corresponds to the worst health you can imagine and score 100 corresponds to the best health you can imagine (collected scores ranged from 10-100). EQ-5D Total Index is based on general population valuation surveys. Responses to 5 questions are converted to an Index value and score range from 0 to 1, with higher scores indicating better quality of life. Total Index was derived on US population (collected scores ranged from 0.4-1). General pain assessment (Pain score) is done through a visual analog scale (VAS), scores ranging from 0 to 100 with higher scores indicating more pain (collected scores ranged 0-87).
Time Frame: Baseline at exposure day 1 and at study completion/termination.
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | BAX 326
Number analyzed (Participants) | 26
Score on a scale
  EQ-5D Total Index | 0.0 (0.13)
  EQ-5D VAS: number analyzed (Participants) | 25
  EQ-5D VAS | 5.1 (21.75)
  Pain Score: number analyzed (Participants) | 24
  Pain Score | -8.0 (36.62)

ADVERSE EVENTS:
Time Frame: Throughout the entire study period from screening to completion/termination. Overall 6 years and 2 months. For each participant the duration of study depended on when the participant has accumulated a total of 100 exposure days during the course of the pivotal/pediatric studies and this study.
Arm/Group | BAX 326
All-Cause Mortality (participants affected / at risk) | 0/115
Serious Adverse Events (participants affected / at risk) | 9/115
Other Adverse Events (participants affected / at risk) | 63/115
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BAX 326 (N=115)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Duodenal ulcer hemorrhage (Gastrointestinal disorders) | 1 (1)
Corneal abscess (Infections and infestations) | 1 (1)
Brain contusion (Injury, poisoning and procedural complications) | 1 (1)
Extradural hematoma (Injury, poisoning and procedural complications) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Scroctal haematoma (Injury, poisoning and procedural complications) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (3)
Renal colic (Renal and urinary disorders) | 2 (3)
Testicular appendage torsion (Reproductive system and breast disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BAX 326 (N=115)
Pyrexia (General disorders) | 14 (23)
Bronchitis (Infections and infestations) | 6 (8)
Influenza (Infections and infestations) | 8 (8)
Nasopharyngitis (Infections and infestations) | 25 (55)
Pharyngitis (Infections and infestations) | 6 (8)
Rhinitis (Infections and infestations) | 8 (15)
Upper respiratory tract infection (Infections and infestations) | 11 (17)
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 (48)
Headache (Nervous system disorders) | 8 (20)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (15)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Hypertension (Vascular disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Agreements may vary with individual PIs, but contain common elements. For this study, PIs are restricted from independently publishing results until the earlier of the primary multicenter publication or up to 2 years after study completion. The sponsor requires a review of results communication (e .g. for confidential information) ≥ 60 days prior to submission and may request an additional delay up to 6 months (e .g. for intellectual property protection). Prior authorization may be required.

DOCUMENTS (2):
  • Study Protocol (2015-10-19): https://cdn.clinicaltrials.gov/large-docs/79/NCT01286779/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-27): https://cdn.clinicaltrials.gov/large-docs/79/NCT01286779/SAP_001.pdf